CLINICAL TRIAL: NCT05836519
Title: The Effect of Pes Planus on Physical Activity Level, Exercise Capacity and Quality of Life in Young Adults
Brief Title: Effects of Pes Planus on Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Meryem Özdemir, Phsiotherapy Student, Saglik Bilimleri Universitesi
Other Study IDs: Effects of Giving Up Planus
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pes Planus
Keywords: Physical Activity; Exercise Capacity; Life Quality
MeSH Terms: conditions — Flatfoot; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with a pes planus: Navicular drop test, International Physical Activity Questionnaire (IPAQ), Digital dynamometer measurement, SF-36 quality of life Questionnaire, 6 Minutes Walk test, Foot Function Index, borg value, heart rate, blood pressure, oxyhemoglobin values will be measured for individuals with pes planus.
  Interventions: Other: Survey Navicular Drop test, International Physical Activity Questionnaire (IPAQ) Short Form, 6-minute walk test, Foot Function Index (AFI), SF-36 quality of life questionnaire, Modified borg scale
- Individuals Without Giving Up Planus: Navicular drop test, International Physical Activity Questionnaire (IPAQ), Digital dynamometer measurement, SF-36 quality of life Questionnaire, 6 Minutes Walk test, Foot Function Index, borg value, heart rate, blood pressure, oxyhemoglobin values will be measured for individuals with pes planus.
  Interventions: Other: Survey Navicular Drop test, International Physical Activity Questionnaire (IPAQ) Short Form, 6-minute walk test, Foot Function Index (AFI), SF-36 quality of life questionnaire, Modified borg scale

INTERVENTIONS:
Other: Survey Navicular Drop test, International Physical Activity Questionnaire (IPAQ) Short Form, 6-minute walk test, Foot Function Index (AFI), SF-36 quality of life questionnaire, Modified borg scale — Pulse oximetry will be used to measure the oxyhemoglobin value of the participants, and a sphygmomanometer will be used for blood pressure and heart rate measurements.
  Other Names: Device Sphygmomanometer, pulseoximeter

SUMMARY:
This study will be conducted to investigate the effect of pes planus on physical activity level, exercise capacity and quality of life in young adults. In the study, various evaluations and questionnaires will be applied to the participants by dividing them into two groups by performing the navicular drop test. In the study, questionnaires and applications such as Digital dynamometer measurements, Foot Function Index (AFI), International Physical Activity Questionnaire (IPAQ), 6 Minute Walk test, blood pressure, heart rate, saturation measurements, Modified Borg Scale and SF-36 quality of life questionnaire will be used.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of pes planus on physical activity level, exercise capacity and quality of life in young adults. There are studies examining the effects of pes planus on physical fitness, quality of life, balance and pain levels. However, there are no studies evaluating the effect of pes planus on exercise capacity and physical activity level. It will enable us to have information about its capacity and its effect on quality of life and to obtain workable data. Thanks to these data, the orientation towards treatment options for the negative effects of pes planus will increase. After the approval of the ethics committee, 32 participants who meet the inclusion criteria will be included in the study. The participants will be divided into two groups, 16 with pes planus and 16 without pes planus, by performing the navicular drop test. The foot muscle strength of the participants will be measured with a digital muscle strength device (Lafayette Manual Muscle). The International Physical Activity Questionnaire (IPAQ) will be used for the physical activity level of the participants, the 6-minute walking test for the exercise capacity, the SF-36 quality of life questionnaire for the quality of life, and the Foot Function Index (AFI) for the foot functional status. Heart rate, blood pressure, borg value and oxyhemoglobin value will be measured before and after the 6-minute walking test to be performed on the participants. According to these measurements, the physical activity levels, exercise capacities and quality of life of the participants in both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30,
* Being able to walk independently (Can use a walking aid)
* Not having a diagnosed psychiatric disorder.

Exclusion Criteria:

* Presence of inflammatory, systemic, degenerative and neurological diseases of the foot and ankle,
* Presence of standing equine, hallux valgus and hallux rigidus deformities
* Current history of surgery related to the foot-ankle,
* Existence of cooperation disorders that would prevent participation in the study.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Young adults aged 18-30 years
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | Baseline
  It will be used to determine whether participants have pes planus. Participants will undergo a navicular drop test to assess arch height, flexibility, and standing pronation. In the sitting position where the participants do not carry weight with bare feet, while their feet are in contact with the ground, a mark will be placed on the card on the floor at the level of the navicular tubercle.
  Then, on the same card, a mark will be made on the same card at the level of the navicular tubercle in the position where they stand up with full weight on the same card. The difference in the distance between the two marked lines will be recorded as the amount of navicular fall in mm. Participants with a diameter of 10 mm or more in the group will be evaluated in the group with pes planus.
Muscle Strength | Baseline
  With the digital muscle strength device, muscle strength assessment will be made on the muscles of the participants who have foot dorsiflexion, plantarflexion, inversion and eversion.
6 minutes walking test | 6 minutes
  The exercise capacity of the participants will be evaluated with the 6-minute walking test.
International Physical Activity Questionnaire-Short form (IPAQ) | Baseline
  The physical activity levels of the participants will be evaluated with the International Physical Activity Questionnaire-Short Form (IPAQ). According to the questions in the questionnaire, metabolic equivalent (MET) scores were determined according to how many days per week, how many hours or minutes per day the activities were performed. According to the survey, it will be determined that as metabolic equivalents increase, physical activity levels are higher, and as they decrease, it will be lower.
Foot Function Index | Baseline
  The foot function status of the participants will be evaluated with the Foot Function Index (AFI). It is a 23-item questionnaire and each item will be given a value between 0-10 according to the visual analog scale and a score will be made between 0-100. The average of all scores will be taken during the calculation. A higher calculated value means more activity limitation, disability, and more pain.
SF-36 quality of life questionnaire | Baseline
  The quality of life of the participants will be evaluated with the Short Form Health Survey (SF-36 Short Form) consisting of 36 questions. This questionnaire evaluates the positive and negative aspects of health status. As a result of the survey, a value between 0-100 will be found. A high score from the scale indicates good quality of life.

SECONDARY OUTCOMES:
Modified Borg Scale | Baseline
  Before and after the 6-minute walk test, the fatigue levels of the participants will be evaluated with the Modified Borg Scale. According to the modified borg scale, participants will score their fatigue with a value between 0 and 10. As the value said by the participants approaches 10, it will be determined that their fatigue levels increase.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, assoc.prof, Study Director — Saglik Bilimleri Universitesi